CLINICAL TRIAL: NCT02388334
Title: Impact of Multiple Sclerosis From the Viewpoint of the Caregivers : Exploring Their Quality Of Life and Their Expectations Concerning the Quality of Professional Management
Brief Title: Impact of Multiple Sclerosis From the Viewpoint of the Caregivers
Acronym: AQUASEP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government); Nantes University Hospital (Other); University Hospital, Angers (Other Government); Central Hospital, Nancy, France (Other); University Hospital, Strasbourg (Other); University Hospital, Marseille (Other); University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: PREPS 13-0227
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Sclerosis
Keywords: Caregivers; Quality of life; Quality of care
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: to develop a standardized questionnaire — to develop, from the caregivers' point of view, a standardized questionnaire evaluating 1) their quality of life (QOL) as related to the disease of the assisted and 2) their expectations concerning the global quality of professional management (care, coordination, information...).
  The development of this standardized tool will also :
  * identify the specific support needs of the caregivers
  * study the links between the quality of care as perceived by the professionals, patients and caregivers
  * identify the characteristics of the caregivers (status) and patients (disease type, disease-modifying drug (DMD) initiation, disease duration) associated with questionnaire results.

SUMMARY:
Half the MS patients require a natural (non professional) caregiver's support for daily living activities and this level of investment increases with the degree of disability.

The caregiver's role is an essential key factor in the "therapeutic alliance" between the patient and heath professionals. The impact on the natural caregivers' Quality Of Life (QOL) and their expectations for the global quality of management are not documented, notably because of the lack of adapted tools.

The aim of the investigators' project is to develop, from the caregivers' point of view, a standardized questionnaire evaluating 1) their QOL as related to the disease of the assisted and 2) their expectations concerning the global quality of professional management (care, coordination, information...).

1) their quality of life (QOL) as related to the disease of the assisted and 2) their expectations concerning the global quality of professional management (care, coordination, information...).

The original tool validated will complete the palette of those that the investigators are developing to evaluate the quality of care of MS patients according to different dedicated organizations (formal networks or not, focused on the patients or professionals).

DETAILED DESCRIPTION:
Half the MS patients require a natural (non professional) caregiver's support for daily living activities and this level of investment increases with the degree of disability. Authors considered that an approach focused on the caregiver's burden limits the perception and evaluation of the real impact of his/her role at the patient's side, just as it probably limits the effectiveness of interventions used and the support they can be offered. According to them, the concept of QOL linked to the disease of the assisted person would be better adapted to respond to this question, because of its multidimensional approach, along with the potential secondary benefits of caregiving.

Although consideration of the patients' point of view to evaluate the effectiveness and quality of therapeutic strategies and, more widely, healthcare interventions have been imposed for the last 20 years in the investigators' healthcare systems, the data on caregivers' viewpoints are more recent. Authors concurred that assessing caregivers' needs and experiences is a more appropriate source of information to identify their expectations concerning the quality of the healthcare system rather than the concept of "patient satisfaction". The impact of MS on the natural caregivers' QOL and expectations for the global quality of management is not documented in France, notably because of the lack of adapted tools. So, if caregivers' support capacities are exceeded primarily because of their own impaired QOL and their expectations for the quality of management are not considered, the therapeutic contract will be diminished, thereby worsening the overall quality of management for MS patients.

The original tool validated will complete the palette of those that the investigators are developing to evaluate the quality of care of MS patients according to different dedicated organizations (formal networks or not, focused on the patients or professionals). All tools will initially be tested together, in the framework of the IRSEP project (funding by the ministry of health : PREQHOS n° 2010-A0096138) on 3 regional population-based cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Age eligible for caregivers and patients : 18 years and over
* Patients with diagnosis of definite MS.
* In order to consider the diversity of the situations, socio-demographics (gender of the patient, status of the caregiver) and disease's evolution (disability status, time since first symptoms) characteristics will be considered for

Exclusion Criteria:

* Caregivers and patients incapable of understanding the proposed procedure and the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Natural caregivers of Multiple Sclerosis patients
Sampling Method: Non-Probability Sample
Enrollment: 730 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Validation phase of the questionnaire | 2 years
  The validation phase of V2 comprises the analysis of the construct's reliability, exploratory and confirmatory stages of tool structuration in dimensions, and the reproducibility of the findings generated. It relies on the recruitment of caregivers who did not participate in the preceding steps.
  To verify the stability of tool responses, another test round by 20% of the responders will be conducted 15 +/- 5 days after the first evaluation.
  Finally, an analysis of sensitivity to change (e.g. initiation of a new treatment, transition to a progressive form; changes in disease management; changes in caregiver's situation) will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: David Veillard, Principal Investigator — Rennes University Hospital